CLINICAL TRIAL: NCT01955148
Title: Prospective Phase III Evaluation Of Fetal Fibronectin In A High Risk Asymptomatic Population For The Prediction Of Spontaneous Preterm Birth
Brief Title: fFN Clinical Evaluation in Asymptomatic Women at High Risk for Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10Q01
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Pre-term Birth
Keywords: PTB; sPTB; cervical cerclage; LEEP; PROM; short cervix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cervicovaginal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prior sPTB or PROM: Women who have had a previous delivery of a live born singleton between 20 weeks, 0 days and 36 weeks, 6 days due to spontaneous preterm premature labor or preterm rupture of fetal membranes
- Short cervical length: Short cervical length (≤25 mm) determined by transvaginal ultrasound
- Twin Pregnancy: Current twin pregnancy
- Prior cervicdal surgeries: Cervical cerclage in a prior pregnancy or prior cone biopsy or prior LEEP

SUMMARY:
This study is designed to determine if quantitative analysis of fetal Fibronectin (fFN) can be used to advance prediction of spontaneous preterm birth (sPTB). This will be a prospective observational multi-center study with approximately 15 to 20 US sites, and approximately 1210 subjects evaluating the clinical utility of the Rapid fFN 10Q system for preterm birth risk assessment. A single fFN specimen will be collected from each subject between 16 weeks, 0 days and 21 weeks, 6 days. The primary and secondary maternal outcome measures will be determined based on the date of delivery and the estimated date of confinement (EDC), which will be evaluated in a standardized manner.

DETAILED DESCRIPTION:
Hologic has developed a quantitative test to assess the amount of fetal fibronectin (fFN) present in cervicovaginal secretions, and evaluate the clinical utility of the test in assessing spontaneous Pre-Term Bith risk in a high risk population. Identifying women at high risk of giving birth prematurely can be challenging. It is believed that higher levels of fFn measured in vaginal fluid suggest a woman is at a greater risk for delivering early. fFN testing is already approved for use in women from weeks 22 to 35 of pregnancy. The goal of this study is to evaluate the benefits of collecting fFN measurements from a vaginal fluid specimen taken during early pregnancy (from 16 weeks to 22 weeks) to assess the risk of pre-term birth.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women from 16 weeks, 0 days to 21 weeks, 6 days' gestation
2. Maternal age ≥18 years of age
3. Subject has signed and dated an Institutional Review Board (IRB) approved consent form to participate in the study
4. Subjects for this study must be at high risk for preterm birth as indicated by at least one of the following:

   * A previous delivery of a live born singleton between 20 weeks, 0 days and 36 weeks, 6 days due to spontaneous preterm premature labor or preterm rupture of fetal membranes
   * Short cervical length (≤25 mm) determined by transvaginal ultrasound
   * Current twin pregnancy
   * Cervical cerclage in a prior pregnancy
   * Prior cone biopsy
   * Prior LEEP / LLETZ

Exclusion Criteria:

1. Maternal age under 18
2. Suspected or proven rupture of fetal membranes at the time of specimen collection
3. Known significant congenital structural or chromosomal fetal anomaly
4. Women with moderate or gross bleeding evident on speculum examination
5. Women who have had sexual intercourse within 24 hours prior to specimen collection
6. Cervical cerclage at time of specimen collection
7. Current triplet (or more) pregnancy
8. Placenta previa with active bleeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only subjects who are at high risk for preterm birth and meet the inclusion criteria will be included in this study. Subjects may be recruited from each clinical site's routine or referral population. Pregnant women who meet the study eligibility criteria will be screened for possible inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1210 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a high and low level of fFN as a Measure of Predicting Pre-Term Birth | 18 months
  To determine whether the rate of spontaneous delivery < 35 weeks in women with a high level of fFN (equivalent to ≥ 200 ng/mL) is greater than in women with a low fFN (< 10 ng/mL) measured from 16 weeks, 0 days to 21 weeks, 6 days' gestation in a high risk coho

SECONDARY OUTCOMES:
Number of Participants with a moderate level of fFN as a Measure of Predicting Pre-Term Birth | 18 months
  To determine whether the rate of spontaneous delivery < 35 weeks in women with a moderate level of fFN (10-199 ng/mL) is greater than in women with a low fFN (< 10 ng/mL) measured from 16 weeks, 0 days to 21 weeks, 6 days' gestation in a high risk cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Sean C Blackwell, MD, Principal Investigator — UTHealth - Medical School at Houston; Errol Norwitz, MD, Ph.D., Principal Investigator — Tufts Medical Center; Joseph Biggio, MD, Principal Investigator — University of Alabama at Birmingham; David Adair, MD, Principal Investigator — Regional Obstetrics Consultants, PC; Anthony Sciscione, MD, Principal Investigator — Christiana Care Health Services, Inc.; Eugene Chang, MD, Principal Investigator — Medical University of South Carolina; Eric Knudtson, MD, Principal Investigator — Board of Regents of the University of Oklahoma; Kathryn Menard, MD, Principal Investigator — University of North Carolina, Chapel Hill; George Saade, MD, Principal Investigator — The University of Texas Medical Branch at Galveston; Catalin Buhimschi, MD, Principal Investigator — Ohio State University; Kira Pryzbylko, MD, Principal Investigator — Lawrence OB/GYN Associates; Glenn Markenson, MD, Principal Investigator — Baystate Medical Center; Hyagriv Simhan, MD, Principal Investigator — University of Pittsburgh - Magee Women's Hospital; Michael S Ruma, MD, Principal Investigator — Perinatal Associates of New Mexico; Allen Rappleye, MD, Principal Investigator — Jean Brown Research
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - Women's Health Care Research Corp., San Diego, California
  - Christiana Hospital, Newark, Delaware
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Lawrence OB/GYN Associates, Lawrenceville, New Jersey
  - Perinatal Associates of New Mexico, Albuquerque, New Mexico
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - University of Texas - Medical Branch at Galveston, Galveston, Texas
  - University of Texas-Houston, Houston, Texas
  - Jean Brown Research, Salt Lake City, Utah